CLINICAL TRIAL: NCT02845830
Title: Trajectories of Quality of Life by the Elderly in Early Phase of Dementia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Palacky University (Other)
Collaborators: University Hospital Ostrava (Other); University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Ing. Irena Jedličková, Study coordinator, Palacky University
Other Study IDs: 16-28628A
Record Dates: First submitted 2016-07-24; First posted 2016-07-27 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Dementia; Quality of Life
Keywords: dementia; elderly; quality of life; assessment; factor; trajectory; change; early stage
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants in early stage of dementia: Subjects with any type of dementia at an early phase diagnosed in the last 12 months with MMSE score 20-25 points
- Participants without dementia: Subjects without dementia with MMSE score 26-30 points

SUMMARY:
Maintaining of improving the quality of life amongst the elderly with early phase dementia (EwD) is nowadays one of the key aims of health care services. When investigating the quality of life trajectories, it is necessary to examine contributing factors. The aim of the project is to ascertain the profile of quality of life trajectory amongst Czech EwD and to identify the most important factors affecting it. The results will be compared to the results from the elderly without dementia. A quantitative approach, longitudinal prospected design utilising a battery of questionnaires in the Czech language will be used. At the same time, translation and validation of the Czech version of QOL-AD and PDI will be carried out. The group of respondents will include EwD and elderly without dementia living in home environment. Knowledge of the quality of life trajectory and the factors involved will enable interventions to maintain or improve the quality of life of the elderly with early-stage dementia in home environment in future. Project Aims The aims are to ascertain the quality of life trajectory profile amongst the elderly with early phase dementia, to identify the most important factors involved and to compare the results to control group. Validation of the Czech versions of QOL-AD and PDI questionnaires will be performed.

DETAILED DESCRIPTION:
Introduction In the Czech Republic, there are about 120 -150 thousand people living with dementia. The most common form of dementia is the Alzheimer's disease, which constitutes about 50 -70 % of all dementia cases and its prevalence in the population is on the rise with the increasing proportion of population over 60 years of age. In 2012, patients with dementia in Alzheimer's disease (AD), who were treated with this disease for the first time, comprised more than 28 % of total number of outpatients treated for dementia. Number of treated patients with dementia increased by 5 % between years 2012 and 2013. According to the World Health Organisation, dementia has become a priority for the health care system. Maintaining or improving the quality of life (QoL) amongst the elderly with dementia is currently one of the key aims of health care. Foreign literature points out the fact that QoL amongst the elderly with dementia (EwD) has not yet been sufficiently examined, particularly in the long-term perspective. This may stem from the fact that QoL amongst the EwD was examined in relation to a relatively limited group of factors. We see an attempt to define each of the factors affecting the quality of life amongst EwD. Among factors with direct impact on the assessment of QoL amongst the EwD is attitude to aging. Social and interpersonal factors also play an important role in the subjective perception of QoL. This includes a decreased ability to communicate which deepens the social isolation at an early-phase dementia, which is reflected negatively in the subjectively perceived QoL amongst EwD. QoL amongst the elderly with slight cognitive impairment and dementia is significantly affected by fear of falling. Other factors include dignity, chronic pain and depression. Another major factor connected with age is frailty, which impairs the ability of the organism to react to stressors and affects QoL. For this reason the relation between frailness and cognitive impairment is studied today. One of the factors affecting QoL amongst EwD is also functional condition. The EwD need an increased amount of supervision and help with activity daily living (ADL) and this dependence negatively affects their QoL. The relation between comorbidity and QoL amongst EwD has not been clearly proved in earlier studies. However, an important aspect of comorbidity is its relation to QoL and health status of the elderly. An early-phase dementia is primarily characterised by memory impairment with a relatively maintained self-sufficiency requiring only minor attention and help by family caregivers. Older adults are usually aware of their condition which may cause depression, anxiety and insecurity. Self-assessment of QoL amongst people with early-phase dementia is supported in the latest research abroad. Cross-sectional studies but a mainly long-term observation of QoL trajectory is important in individuals with dementia. When investigating the trajectory of QoL amongst EwD, it is necessary to examine the factors which might affect QoL. So far, there have been few longitudinal studies focusing on changes in QoL in connection with progressing dementia and contributing factors. This may be due to the fact that the QoL amongst EwD was examined in relation to a relatively limited group of factors, even though previous research recommended to examine the changes in QoL amongst EwD in the long run and in a larger group of respondents.

Project Objectives In order to maintain the maximum possible quality of life in people suffering from a disease of the nervous system, an early diagnosis and therapy is necessary, as well as nursing and psychosocial care.

The aim is not only to improve the quality of life with a lower frequency and length of hospitalisations, but also to enhance individual's resilience.

The chance to express the quality of life subjectively shifts the assessment of health care results from a solely medical perspective to an assessment from the perspective of a concrete individual.

The objective of the project is a monitoring of the trajectory of subjectively perceived quality of life amongst the elderly with early-phase dementia in the long run. Identifying the factors and their effect on the quality of life may help to enhance resilience of the elderly and to have a positive effect on the physical, psychosocial and social dimension of the quality of life with early-phase dementia in home care and thus lower the frequency and length of hospitalisations as well as costs in health care and social care.

The main aim of the project is to ascertain how quality of life changes amongst Czech elderly with early-phase dementia (quality of life trajectory). To achieve the main aim, five sub-aims have been set, which should support the investigation of quality of life in patients with a nervous system disease, namely amongst the elderly at an early phase of dementia.

1. Translation and validation of Czech versions of standardised QOL-AD and PDI questionnaires.
2. Identification of the most important factors contributing to the changes in quality of life among Czech elderly with early-phase dementia.
3. Creation of a profile of quality of life trajectory amongst Czech elderly at an early phase of dementia.
4. Comparison of the trajectory of Czech elderly with early-phase dementia to the trajectory of the elderly not diagnosed with dementia.
5. Creation of a database for subsequent longitudinal trajectory tracking the quality of life of older people with dementia Methodology In order to achieve the goals of the project, a prospective, longitudinal design using quantitative method will be used - a survey research will be carried out in a group of respondents on entering the study and repeated twice subsequently at 12-month interval.

Prior to the 1st stage of the survey research, a translation and validation of QOL-AD and PDI questionnaires will be done. Based on the results of international studies, a group of factors was identified which affect quality of life in the elderly with dementia.

The research will be carried out using a batch of standardised Czech versions of questionnaires related to these factors: Quality of Life - Alzheimer's Disease (QOL-AD); Geriatric Depression Scale by Yesavage (GDS-15) - Czech version; Mini Mental State Exam (MMSE - Czech version). In case the use of MMSE is bound with licence fees a Czech version of the Addenbrook Cognitive Examination (ACE-CZ) will be used; Patient Dignity Inventory (PDI); Attitude to Aging Questionnaire (AAQ) - Czech version; Falls Efficacy Scale International (FES-I) - Czech version; Short Physical Performance Battery (SPPB) - Frail Index; Bristol Activities of Daily Living Scale (BADLS-CZ), Horizontal visual analog scale (HVAS). Furthermore, the comorbidity index and basic demographic data (age, sex, socio-economic status, education) will be gathered and evaluated.

Research sample will consist of two groups of older adults. The first (patient) group: elderly with a diagnosed dementia at an early phase (F00, F01-F03) will be addressed together with their family caregivers via neurologic outpatient offices, where the elderly are treated for the diagnoses.

The second (control) group: elderly without dementia, addressed through GP's surgeries.

The respondents will be gathered in the Olomouc, Moravia-Silesia and Hradec Králové Regions. Sample size: 580 respondents (290 older adults with dementia and 290 older adults without dementia).

ELIGIBILITY:
Inclusion Criteria:

age ≥60 years lives at home MMSE 20 - 30 points contact with a family caregiver (if any) at least once a week who gives consent to be included in the survey

Exclusion Criteria:

severe psychic disorder severe sensory impairment (vision, hearing) long-term residence in a facility (care home)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly aged ≥60 years
Sampling Method: Non-Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-01 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Quality of Life - Alzheimer's Disease (QOL-AD) | 24 month
  Quality of life questionnaire

SECONDARY OUTCOMES:
Geriatric Depression Scale by Yesavage (GDS-15) | 24 month
  Depression questionnaire
Mini Mental State Exam (MMSE) | 24 month
  Cognitive function questionnaire
Patient Dignity Inventory (PDI) | 24 month
  Dignity questionnaire
Attitude to Aging Questionnaire (AAQ) | 24 month
  Attitude to aging questionnaire

OTHER OUTCOMES:
Falls Efficacy Scale International (FES-I) | 24 month
  Falls efficacy questionnaire
Short Physical Performance Battery (SPPB) - Frail Index | 24 month
  Physical performance questionnaire
Bristol Activities of Daily Living Scale (BADLS-CZ) | 24 month
  Activities of daily living questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Helena Kisvetrova, PhD, Principal Investigator — Faculty of Health Science, Palacký University Olomouc

IPD SHARING:
Plan to Share IPD: Undecided